CLINICAL TRIAL: NCT05952934
Title: A Phase II Clinical Trial of Candida Therapeutic Vaccine in Head and Neck Cancer Patients to Reduce Recurrence
Brief Title: Candida Therapeutic Vaccine in Head and Neck Cancer Patients to Reduce Recurrence
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Arkansas (Other)
Collaborators: Highlands Oncology Group, PA (Unknown); NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 275695
Record Dates: First submitted 2023-07-03; First posted 2023-07-19 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Squamous Cell Carcinoma of Head and Neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: This is a Phase II randomized, double-blind, placebo controlled, multi-site study of Candin.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Each study site will received a separate randomization scheme, and the research pharmacy at each site will implement and maintain randomization schedule.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Candin vaccine (Active Comparator): Seven Candida (Candin). The route of administration is intradermal injection at subject's limbs at 0.5 mL/injection. The schedule is 1 injection every three weeks for the first 4 injections, and then one injection every 3 months until a total of 7 injections has been given.
  Interventions: Biological: 0.5 mL Candin®/injection
- Placebo (Placebo Comparator): Seven placebo injections (sterile 0.9% Normal Saline). The route of administration is intradermal injection at subject's limbs at 0.5 mL/injection. The schedule is 1 injection every three weeks for the first 4 injections, and then one injection every 3 months until a total of 7 injections has been given.
  Interventions: Other: Placebo: 0.5 mL Intravenous 0.9% NaCl solution (Saline)

INTERVENTIONS:
Biological: 0.5 mL Candin®/injection — Candin or placebo injection every 3 weeks until 4 injections then every 3 months until a total of 7 injections.
  Arms: Candin vaccine
Other: Placebo: 0.5 mL Intravenous 0.9% NaCl solution (Saline) — Placebo injection every 3 weeks until 4 injections then every 3 months until a total of 7 injections.
  Arms: Placebo

SUMMARY:
This is a Phase II randomized, double-blind, placebo controlled, multi-site study of Candin. It is designed to show the efficacy and safety of a 7-dose regimen of Candin over a two-year period in terms of reducing cancer recurrence rate by comparing the recurrence rates between the Candin and the placebo arm. The ratio of the number of subjects who will receive Candin versus placebo will be 3:1. Up to 100 subjects will be screened until 80 subjects are eligible for injection.

DETAILED DESCRIPTION:
This is a Phase II study to evaluate the efficacy and safety of a therapeutic vaccine called Candin® (Nielsen Biosciences, San Diego, CA) in adults over a two (2) year period. Each subject will be receiving a total of 7 injections of Candin (0.5 mL per dose) or placebo (saline) at a 3:1 ratio in a randomized double-blinded design. Subjects will receive one injection every 3 weeks until they receive 4 injections. Then, subjects will receive one injection every 3 months until they receive a total of 7 injections. Subjects will have 2 more visits approximately 6 months apart after the last injection. Immunological assessment T-cell repertoire analysis and by fluorescent activated cell sorter analysis (FACS) will be made at 4 time points (Visits 1, 5, 7, and 8). Stool and oral wash samples will be collected at the Screening Visit, Visit 5, Visit 7 and Visit 8 for microbiome diversity analysis.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent
* Male or female 18 years of age or older
* Squamous cell carcinoma of the head and neck who have completed curative therapy (surgery and/or radiation and/or chemotherapy) within the previous 120 days.
* No Evidence of Disease (NED) based on clinical and/or radiographic evaluations
* Willing and able to comply with the requirements of the protocol

Exclusion Criteria:

* Positive urine pregnancy test for women of childbearing potential
* Being pregnant or attempting to be pregnant with the period of study participation
* Women who are breast feeding or plan to breast feed within the period of study participation
* Patients who are allergic to Candin®
* If in the opinion of the PIs or other Investigators, it is not in the best interest of the patient to enter or continue in this study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-02-12 (Actual); Primary Completion 2029-02-01 (Estimated); Study Completion 2029-02-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of clinical efficacy | Through study completion, up to 2 years
  Studying the efficacy of Candida and the schedule in which this protocol specifically outlines the clinical response (i.e., reduced cancer recurrence rate) of subjects is the primary endpoint.

SECONDARY OUTCOMES:
Assessment of adverse events | Regularly throughout the study, up to 2 years
  The secondary endpoints of this study is safety, and the AEs will be diligently recorded and reviewed.

CONTACTS AND LOCATIONS:
Overall Officials: Omar Atiq, Principal Investigator — University of Arkansas
Locations (6):
- United States (6):
  - Highlands Oncology Group, PA, Fayetteville, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Highlands Oncology Group, PA, Rogers, Arkansas
  - Highlands Oncology Group, PA, Springdale, Arkansas
  - Perlmutter Cancer Center at NYU Langone Health, Mineola, New York
  - Perlmutter Cancer Center at NYU Langone Health, New York, New York